CLINICAL TRIAL: NCT07101276
Title: Effect of Core Muscle Endurance on Punch Speed and Force in Boxers
Status: Completed | Type: Observational
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Mehmet Miçooğulları, Asst. Prof. Dr., Cyprus International University
Other Study IDs: 020-4522
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Sports Physical Therapy
Keywords: Core Muscle; Endurance; Punch speed; Boxer; Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Licensed Boxers: Highly trained licensed boxers from a national team in North Cyprus
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be performed in this study.

SUMMARY:
This cross-sectional within-subject design study aimed to investigate the contribution of core muscles to punch speed and power among highly trained licensed boxers from a national team in North Cyprus.

DETAILED DESCRIPTION:
From a biomechanical point of view, the high-impact force generated by the lower limbs in boxers is transferred through the stiff kinetic chain, which is stabilised by the core muscles to transform into a powerful punch in the upper extremity. Despite these essential functions, there is a lack of research on the effect of core muscles in boxing. Therefore, this study aimed to investigate the contribution of core muscles in punching, and it was hypothesised that the endurance of trunk flexors, extensors, and lateral muscles on the dominant and non-dominant sides has a substantial contribution to punch speed and power in boxers.

ELIGIBILITY:
Inclusion Criteria:

* Licensed boxers aged 18-35 years
* Free of injuries
* No history of surgery, visual, or vestibular disorders

Exclusion Criteria:

* Presence of any injury
* History of surgery, visual, or vestibular disorders
* Outside the age range of 18-35 years
* Not holding a valid boxing license

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Licensed boxers from a national team in North Cyprus
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Endurance of trunk flexor muscles | 1 hour
  The athlete will be positioned on a flat surface. The tester will stabilise the feet while the hip and knee joints are placed at 90 degrees of flexion. The upper extremities will be crossed over the shoulders, bringing the trunk into approximately 60-degree flexion.
Endurance of trunk extensor muscles | 1 hour
  Subjects will lie prone with the lower body fixed to the test bed at the ankles, knees, and hips, and the upper body extended in a cantilevered fashion over the edge of the test bed. At the beginning of the exertion, the upper limbs will be held across the chest with the hands resting on the opposite shoulders, and the upper body will be lifted until the thoracic region is horizontal to the floor.
Endurance of Lateral Trunk (Oblique) Muscles | 1 hour
  Subjects will lie on an exercise mat on their sides with legs extended. The top foot will be placed in front of the lower foot on the mat for support. Subjects will be instructed to support themselves by lifting their hips off the mat to maintain a straight line over their whole body length, and support themselves on one elbow and their feet. The uninvolved arm will be held across the chest with the hand placed on the opposite shoulder.
Evaluation of Punch Speed and Power | 1 hour
  The rear direct punch type will be selected for the test. Punch speed and power will be tested using the Corner Accelerometer (Corner Wearables Ltd / UK), which has been found suitable for tracking punches. The devices will be fixed to both wrists of the boxers with Velcro and paired with the Corner mobile app via Bluetooth. Subjects will perform three rounds of shadow boxing using standard boxing gloves, with five minutes of rest between rounds for warm-up and device checking. Finally, the athletes will be asked to throw a total of five rear direct punches to the boxing bag using their dominant side, and the device will record the parameters of each punch separately and simultaneously, including speed in meters per second (m/sec) and power in gravitational force units (G-force). Of the five punches thrown, the fastest and most powerful will be selected for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Angın, Prof. Dr., Study Director — Cyprus International University
Locations (1):
- Cyprus International University, Mersin, Lefkosa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Dunn EC, Humberstone CE, Franchini E, Iredale KF, Blazevich AJ. Relationships Between Punch Impact Force and Upper- and Lower-Body Muscular Strength and Power in Highly Trained Amateur Boxers. J Strength Cond Res. 2022 Apr 1;36(4):1019-1025. doi: 10.1519/JSC.0000000000003585. PMID 32218063
- [Background] Rodriguez-Perea A, Reyes-Ferrada W, Jerez-Mayorga D, Chirosa Rios L, Van den Tillar R, Chirosa Rios I, Martinez-Garcia D. Core training and performance: a systematic review with meta-analysis. Biol Sport. 2023 Oct;40(4):975-992. doi: 10.5114/biolsport.2023.123319. Epub 2023 Feb 3. PMID 37867742
- [Background] Shinkle J, Nesser TW, Demchak TJ, McMannus DM. Effect of core strength on the measure of power in the extremities. J Strength Cond Res. 2012 Feb;26(2):373-80. doi: 10.1519/JSC.0b013e31822600e5. PMID 22228111
- [Background] Akuthota V, Nadler SF. Core strengthening. Arch Phys Med Rehabil. 2004 Mar;85(3 Suppl 1):S86-92. doi: 10.1053/j.apmr.2003.12.005. PMID 15034861
- [Background] Beattie K, Ruddock AD. The Role of Strength on Punch Impact Force in Boxing. J Strength Cond Res. 2022 Oct 1;36(10):2957-2969. doi: 10.1519/JSC.0000000000004252. Epub 2022 Jul 8. PMID 35836314